CLINICAL TRIAL: NCT06270420
Title: Treatment Improvement With the Use of Innovative Technologies and Robotics in Rehabilitation Process: Observational Longitudinal Pilot Study
Brief Title: Technological Devices and Home Automation System in Neurological Rehabilitation
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022.04
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Neurological Disease; Motor Disorders
Keywords: Home Automation; Sensorized environment; Organizational model; Neurological rehabilitation; Technological Innovation; Motor Recovery
MeSH Terms: conditions — Nervous System Diseases; Motor Disorders

STUDY DESIGN:
Intervention Model Description: Longitudinal Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HosmartAI training (Experimental): HosmartAI training will consist of motor training provided by technological devices (i.e. OAK, VRRS, AMADEO, PABLO) in the HoSmartAI room.
  Interventions: Device: Technological Motor Rehabilitation

INTERVENTIONS:
Device: Technological Motor Rehabilitation — Patients will undergo to motor treatment in the HoSmartAI room using one of the technological devices (i.e. OAK, VRRS Evo by Khymeia Group, Padova, Italy; AMADEO, PABLO by Tyromotion GmbH, Gratz, Austria), for the upper limb and lower limb motor recovery, balance and manual dexterity recovery. The duration of the treatment will be 15 sessions, 1 hour each, with daily frequency, 5 days a week, for a total of 3 weeks.

SUMMARY:
The use of home automation system may be useful in rehabilitation to collect data about the environment and the amount of therapy. Then, the data may be stored in a cloud and integrated with data collected during training provided by technological devices.

The main goal of this longitudinal pilot study is to define the productivity of the rehabilitation room (i.e., HoSmartAI room) in the IRCCS San Camillo Hospital (Venice, Italy) service, where the investigators will install home automation sensors and treat patients with neurological disease using technological devices (e.g., robotic and virtual reality). The secondary goals are to define the patients' satisfaction, usability of the system and the clinical effect of treatments delivered with technological devices in the HoSmartAI room. The patient will be assessed to personalized the treatment based on their needs. The treatment will consist of 15 sessions (1h/day, 5day/week, 3 weeks). At the end of the study, the patients will be assessed to define any clinical improvements. Finally, the investigators will define the characteristics of the patients who will benefit from the rehabilitation provided in the HoSmartAI room.

DETAILED DESCRIPTION:
The recovery of motor function is a primary goal for individuals diagnosed with neurological disease, such as Stroke, Parkinson's Disease, Multiple Sclerosis. Various rehabilitation methods have been using in neurorehabilitation hospital, including conventional training and those involving technological devices. Nowadays, the integration of technology into rehabilitation room has been expanding within the National Health System, and their effectiveness in enhancing functionality and quality of life remains a subject of ongoing research in rehabilitation. In addition to rehabilitation devices, such as robotic and virtual reality systems, home automation system may play a crucial role in monitoring and recording patient movements. These sensors can also be employed for home automation in environments such as hospital rehabilitation settings, helping to reduce paid carer hours, quantify the impact of automated data acquisition on the functionality and offer many benefits to people with a disability. Indeed, potentially, the application of home automation system in technological rehabilitation rooms, may allow for the synchronization of environmental data with the patient's clinical history, facilitating the study of functional recovery.

This study is a part of the HosmartAI project (EU Horizon 2020 research and innovation program - grant agreement No 101016834 Pilot #3). The main aim of HoSmartAI project is to develop hospitals based on artificial intelligence (AI) technologies. In Pilot #3, the investigators will integrate data collected by technological devices for motor rehabilitation and home automation sensors installed in room (HosmartAI room) at the Neuromotor Rehabilitation Service of the San Camillo IRCCS Hospital (Venice, Italy). These sensors are able to detect the effective numbers of minutes of therapy, the number of sessions delivered in the room, and detect the presence and falls of the patients. Moreover, all these sensors are managed directly by physiotherapists through an App for smartphone. All data collected will be integrated in a cloud infrastructure, where physiotherapist will check the patients' profile and data collected from clinical assessment and home automation sensors.

In the study, the investigators will enroll patients with neurological disease and motor impairment who are hospitalized in Camillo IRCCS Hospital (Venice, Italy). The treatment (5time/week, for 3 weeks) will consist of 1 hour/day of motor training provided by technological devices (i.e., OAK, VRRS, AMADEO, PABLO) in the HoSmartAI room, in addition to daily 1 hour of conventional motor training. Firstly, the patients will be assessed to define their motor function and personalize the treatment based on their needs, to improve balance, manual dexterity, or upper and lower limb motor recovery. Then, at the end of the treatment, the patients will be assessed using validated clinical scales and questionnaire to determine the clinical effect and patient-reported outcome measurements (i.e., usability, technology acceptability, and user satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 yy)
* Diagnosis of neurological disease (e.g. ischemic and/or hemorrhagic stroke, Parkinson's, multiple sclerosis, brain trauma, peripheral neuropathy)

Exclusion Criteria:

* Fractures
* Major depressive disorder
* Severe visual and/or hearing impairments
* Dementia
* Non-pharmacologically controlled epilepsy
* Severe neglect
* Severe comprehension deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Key performance indicator (KPI) of the room - Number of treatments | Every month up to 1 year
  Number of treatments that are provided inside the HoSmartAI room.
Key performance indicator (KPI) ot the room - Number of sessions | Every month up to 1 year
  Number of sessions that are provided inside the HoSmartAI room.
Room Key performance indicator (KPI) of the room - Number of minutes of therapy | Every month up to 1 year
  Number of minutes of therapy that are provided inside the HoSmartAI room.
Key performance indicator (KPI) of the room - Number of physiotherapists involved | Every month up to 1 year
  Number of physiotherapists involved inside the HoSmartAI room.
Key performance indicator (KPI) of the room - Number of adverse events | Every month up to 1 year
  Number of adverse events detected in the HoSmartAI room.

SECONDARY OUTCOMES:
Box and Blocks Test | Change from Baseline Box and Blocks Test at 3 weeks
  The patient has to carry as much cubes as possible, one by one, from a box to another one in one minute. The test is performed with both hands.
Reaching Performance Scale | Change from Baseline Reaching Performance Scale at 3 weeks
  Reaching Performance Scale assesses the ability of subjects to reach an object (acone). The cone is placed at both 4-cm (close) and 30-cm (far) distance from the subject. The subject is asked to reach and grab the cone if possible. The assessor valuates the quality of reaching instead of the grip strength. The minimum value is0 points, which corresponds to incapacity of any ability of reaching an object. The maximum value is 36 points, which corresponds to the preservation of the ability to reach an object.
Nine Hole Pegboard Test | Change from Baseline Nine Hole Pegboard Test at 3 weeks
  Nine Hole Pegboard Test measures the dexterity of the hand. Patient should insert 9 pins in the board. The number of pins inserted in 50 sec are registered or if the patient inserted 9 pins, then the time is registered.
Berg balance scale (BBS) | Change from Baseline BBS at 3 weeks
  BBS is a 14-item objective measure that assesses static balance and fall risk in adults. The minimum value is 0 (i.e., no stability and high fall risk) and the maximum value is 56 (i.e., no balance disorder and no fall risk).
10 Meter Walk Test (10MWT) | Change from Baseline 10MWT at 3 weeks
  The 10MWT assesses walking speed in meters per second over a short duration.The individual is instructed to walk a set distance (6 meters, 10 meters, etc). Time is measured while the individual walks the set distance (often the individual is given space to accelerate to his/her preferred walking speed (this distance is not included when determining speed). The distance covered is divided by the time it took the individual to walk that distance.Assistive devices may be used but must be documented from test to test.If a patient requires assistance, only the minimum amount of assistance required for a patient to complete the task should be provided. The level of assistance documented, however, should reflect the greatest amount of assistance provided during the test.
Functional Ambulation Categories (FAC) | Change from Baseline FAC at 3 weeks
  FAC is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. The minimum value is 0 (i.e., patient cannot walk) and the maximum value is 6 (i.e., patient can walk independently anywhere).
Trunk Control Test (TCT) | Change from Baseline TCT at 3 weeks
  The TCT measures four simple aspects of trunk movement :rolling to weak side,rolling to strong side
  * balance in sitting position
  * sit up from lying down
EuroQol questionnaire (EQ-5D) | Change from Baseline EQ-5D at 3 weeks
  EQ-5D is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems."
System Usability Scale (SUS) | Change from Baseline SUS at 3 weeks
  SUS is a widely used questionnaire for assessing the perceived usability of a system or product.The SUS consists of a 10-item questionnaire where users rate their agreement or disagreement with a series of statements regarding the usability of a system. The minimum value is 0 (i.e., the system is not usable) and the maximum value is 100 (i.e., the system is absolutely usable).
Short Form Patient Satisfaction Questionnaire (PSQ-18) | Change from Baseline PSQ-18 at 3 weeks
  he Patient Satisfaction Questionnaire Short Form (PSQ-18) is a validated tool used to measure patient satisfaction with medical care. It is a shorter version of the 50-item Patient Satisfaction Questionnaire III (PSQ-III) 1. The PSQ-18 contains 18 items that measure seven dimensions of satisfaction with medical care: general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, and accessibility and convenience
User Experience Questionnaire (UEQ) | Change from Baseline UEQ at 3 weeks
  UEQ is a widely used questionnaire to measure the subjective impression of users towards the user experience of products. The UEQ is a semantic differential with 26 items that are grouped into six scales (Attractiveness, Perspicuity, Efficiency, Dependability, Stimulation, and Novelty). Each scale represents a distinct UX quality aspect. The minimum value is 0 (i.e., the worst user experience) and the maximum value is 100 (i.e., the best user experience).
Number of falls | Require multiple time points before the training to obtain the value (i.e.,12 months, 3 weeks)
  The patients has to count the number of falls in the last year (i.e., 12 months) and in the last 3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgia Pregnolato, Study Chair — IRCCS San Camillo Hospital
Locations (1):
- IRCCS San Camillo Hospital, Venice-Lido, Venice, Italy

REFERENCES:
- [Background] Molteni F, Gasperini G, Cannaviello G, Guanziroli E. Exoskeleton and End-Effector Robots for Upper and Lower Limbs Rehabilitation: Narrative Review. PM R. 2018 Sep;10(9 Suppl 2):S174-S188. doi: 10.1016/j.pmrj.2018.06.005. PMID 30269804
- [Background] Orihuela-Espina F, Roldan GF, Sanchez-Villavicencio I, Palafox L, Leder R, Sucar LE, Hernandez-Franco J. Robot training for hand motor recovery in subacute stroke patients: A randomized controlled trial. J Hand Ther. 2016 Jan-Mar;29(1):51-7; quiz 57. doi: 10.1016/j.jht.2015.11.006. Epub 2015 Nov 26. PMID 26847320
- [Background] Latella D, Maggio MG, Maresca G, Andaloro A, Anchesi S, Pajno V, De Luca R, Di Lorenzo G, Manuli A, Calabro RS. Effects of domotics on cognitive, social and personal functioning in patients with Parkinson's disease: A pilot study. Assist Technol. 2022 Jul 4;34(4):423-428. doi: 10.1080/10400435.2020.1846095. Epub 2021 Apr 6. PMID 33337294
- [Background] Maggio MG, Maresca G, Russo M, Stagnitti MC, Anchesi S, Casella C, Zichitella C, Manuli A, De Cola MC, De Luca R, Calabro RS. Effects of domotics on cognitive, social and personal functioning in patients with chronic stroke: A pilot study. Disabil Health J. 2020 Jan;13(1):100838. doi: 10.1016/j.dhjo.2019.100838. Epub 2019 Sep 4. PMID 31501039
- [Background] Wolbring G, Lashewicz B. Home care technology through an ability expectation lens. J Med Internet Res. 2014 Jun 20;16(6):e155. doi: 10.2196/jmir.3135. PMID 24956581
- [Background] Cleland J, Hutchinson C, Williams PAH, Manuel K, Laver K. A scoping review to explore the health, social and economic outcomes of home automation for people with disability. Disabil Rehabil Assist Technol. 2024 May;19(4):1446-1453. doi: 10.1080/17483107.2023.2196308. Epub 2023 Apr 3. PMID 37012673
- See also: The link of the Pilot #3 refers to the HoSmartAI projects — https://www.hosmartai.eu/pilots/pilot-3/